CLINICAL TRIAL: NCT02929498
Title: A Phase I/II, Open-label, 2 Arm Study to Investigate the Safety, Clinical Activity, Pharmacokinetics and Pharmacodynamics of GSK2879552 Administered Alone or in Combination With Azacitidine, in Adult Subjects With IPSS-R High and Very High Risk Myelodysplastic Syndromes (MDS) Previously Treated With Hypomethylating Agents (HMA)
Brief Title: Safety, Clinical Activity, Pharmacokinetics (PK) and Pharmacodynamics Study of GSK2879552, Alone or With Azacitidine, in Subjects With High Risk Myelodysplastic Syndromes (MDS)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The risk benefit in the study population does not favor continuation of the study
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205744; 2016-002294-35 (EudraCT Number)
Record Dates: First submitted 2016-09-27; First posted 2016-10-11 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Myelodysplastic Syndrome; Myelodysplastic Syndromes
Keywords: GSK2879552; Revised International Prognostic Scoring System (IPSS-R); azacitidine; hypomethylating agents; myelodysplastic syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — GSK2879552; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: GSK2879552 monotherapy (Experimental): Subjects will receive GSK2879552 2 milligrams (mg) once daily in each 28 day cycle.
  Interventions: Drug: GSK2879552
- Arm B: GSK2879552+Azacitidine combination therapy (Experimental): Subjects will receive GSK2879552 starting at 1 mg once daily in each 28 day cycle and Azacitidine 75 mg/square meter (m2) from Day 1 to Day 7 of each 28 day cycle.
  Interventions: Drug: GSK2879552; Drug: Azacitidine

INTERVENTIONS:
Drug: GSK2879552 — GSK2879552 will be administered orally as continuous daily dosing.
Drug: Azacitidine — Azacitidine will be administered at 75 mg/m2 from Day 1 to Day 7 of each 28 day cycle by intravenous (iv) infusion or subcutaneous (sc) injection.
  Arms: Arm B: GSK2879552+Azacitidine combination therapy

SUMMARY:
This is a Phase I/II, open-label, 2 arm study to evaluate the safety and clinical activity of GSK2879552 alone, or in combination with azacitidine in subjects with MDS. The study consisted of 2 parts. The objective of Part 1 is to determine the recommended phase 2 dose (RP2D) of GSK2879552 administered alone and in combination with azacitidine in adult subjects with high risk MDS previously treated with HMA. The objective of Part 2 is to evaluate clinical activity after treatment with GSK2879552, alone or in combination with azacitidine, in adult subjects with high risk MDS previously treated with HMA.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age and provided signed written informed consent
* Subjects must have IPSS-R high or very high risk myelodysplastic syndromes (MDS) by World Health Organization (WHO) classification
* Subjects must have failed hypomethylating treatment where "failure" is defined as: Progression (according to 2006 International Working Group [IWG] criteria) at any time after initiation of the hypomethylating treatment OR Failure to achieve complete or partial response or hematological improvement (HI) (according to 2006 IWG) after at least 4 cycles treatment OR Relapse after initial complete or partial response or HI (according to 2006 IWG criteria).
* Subjects are not a candidate, or have failed allogeneic stem cell transplantation. Subjects who underwent allo-transplant in the past are eligible under following conditions: transplant was >2 year prior to enrolment, and no evidence of active graft-versus-host disease (GVHD)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Subjects must have a life expectancy of at least 12 weeks, in the opinion of the investigator.
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* All prior treatment-related toxicities must be National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 4.0 <=Grade 1 at the time of enrollment (except for alopecia).
* Adequate baseline organ function defined by: International Normalization Ratio (INR) and activated partial thromboplastin time (aPTT) <=1.3xupper limit of normal (ULN); platelet count (PLT) >=10,000 (transfusions permitted to bring PLT to >10,000); total bilirubin <=1.5xULN (Isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35% or subject has a diagnosis of Gilbert's syndrome); Alanine transaminase (ALT) <=2.5xULN; creatinine <=1.5xULN OR calculated creatinine clearance by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation or measured from 24 hour urine >=50 milliliters (mL)/minute (min); and Ejection fraction >=lower limit of normal (LLN) by Echocardiogram (ECHO) or multigated acquisition scan (MUGA)
* Women of childbearing potential must have a negative serum pregnancy test within 7 days of first dose of study treatment and agree to use effective contraception during the study and for 7 days following the last dose of study treatment.
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from the administration of the first dose of study treatment until 3 months after the last dose of study treatment to allow for clearance of any altered sperm.

Exclusion Criteria:

* AML according to world health organization (WHO) criteria (i.e. bone marrow blasts >20%)
* Active hepatitis B or hepatitis C treatment
* Baseline Montreal Cognitive Assessment (MOCA) score of 22 or lower
* History of or concurrent malignancy of solid tumours, except for below:

Exception: Subjects who have been disease-free for 2 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.

* Prior treatment with temozolomide, dacarbazine or procarbazine
* Prior treatment with poly adenosine diphosphate (ADP) ribose polymerase (PARP) inhibitors (example (e.g.), olaparib, veliparib [ABT-888])
* Currently receiving other anti-cancer therapy (chemotherapy, radiation therapy, immuno- therapy, biologic therapy, hormonal therapy, surgery, and/or tumour embolization)
* Received major surgery, radiotherapy, or immunotherapy within 4 weeks of GSK2879552 administration
* Evidence of severe or uncontrolled systemic diseases (e.g., severe/chronic infection, unstable or uncompensated respiratory, renal, or cardiac disease). Any serious and/or unstable pre-existing medical (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator's assessment)
* Patients with any major bleeding current or within the past 4 weeks. (e.g. recent gastrointestinal [GI] hemorrhage or neurosurgery).
* Administration of an investigational drug within 14 days or 5 half-lives, whichever is shorter, preceding the first dose of study treatment(s) in this study.
* Cardiac abnormalities as evidenced by any of the following: clinically significant uncontrolled arrhythmias or uncontrolled hypertension; history or evidence of current >=Class II congestive heart failure as defined by New York Heart Association (NYHA); history of acute coronary syndromes (including unstable angina and myocardial infarction), coronary angioplasty, or stenting within the past 3 months; baseline Corrected QT (QTc) interval using Fridericia's formula >450 milliseconds (msec) or >480 msec in subjects with Bundle Branch Block. QTc value based on single or average of triplicate ECGs obtained over a brief recording period
* Current use of a prohibited medication including anticoagulants or platelet inhibitors or expected to require any of these medications during treatment with the investigational drug
* Consumption of Seville oranges, grapefruit, grapefruit hybrids, grapefruit juice, pommelos, or exotic citrus fruits, from 1 day prior to the first dose of study treatment(s) until the last dose of study drug
* Lactating female
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to GSK2879552 or lysine-specific demethylase 1 (LSD1) inhibitors that contraindicates their participation
* Known hypersensitivity to azacitidine or mannitol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (4):
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Houston, Texas
- Spain (2):
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, 2 arm study to evaluate the safety and clinical activity of GSK2879552 alone, or in combination with azacitidine in adult participants with myelodysplastic syndromes (MDS). The study was conducted in 3 centers among 2 countries.
Pre-assignment Details: Total 5 participants were included into Part 1 and received GSK2879552. The study was terminated during Part 1 and hence Part 2 was not conducted as the risk benefit in earlier studies do not favor continuation of this study.
Groups:
- Part 1: GSK2879552; Part 2: GSK2879552: Participants in this monotherapy arm were administered with GSK2879552 0.5 milligrams or 2 milligrams oral capsules once a day as continuous daily dosing in each cycle (of 28 days) until disease progression during Part 1 of the study.
- Part 2: GSK2879552+Azacitidine: Part 2 was to be initiated once Part 1 is completed and dose has been selected for GSK2879552 monotherapy and combination of azacitidine with GSK2879552. Treatment with GSK2879552 in this combination therapy arm was to be administered orally once a day at RP2D as continuous daily dosing in each cycle (of 28 days) until disease progression in Part 2 of the study. Azacitidine was to be administered at 75 milligram per meter^2 on Days 1-7 of each 28 day cycle by intravenous (IV) infusion or subcutaneous (SC) injection (route of administration: by physicians choice).
Period: Part 1: Dose Confirmation (Upto 2 Years)
Arm/Group | Part 1: GSK2879552 | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Started | 5 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 5 | 0 | 0
Not completed — Study terminated by sponsor | 3 | 0 | 0
Not completed — Death | 2 | 0 | 0
Period: Part 2 : Dose Expansion (Upto 2.5 Years)
Arm/Group | Part 1: GSK2879552 | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part 1 data is presented as study was terminated during Part 1 and hence Part 2 was not initiated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: GSK2879552 | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine | Total
Number analyzed (Participants) | 5 | 0 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] — Part 1 data is presented as study was terminated during Part 1 and hence Part 2 was not initiated.
  Years | 77.2 (5.07) |  |  | 77.2 (5.07)
Sex: Female, Male [Count of Participants; unit: Participants] — Part 1 data is presented as study was terminated during Part 1 and hence Part 2 was not initiated.
  Participants
    Female | 3 | 0 | 0 | 3
    Male | 2 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Part 1 data is presented as study was terminated during Part 1 and hence Part 2 was not initiated.
  Participants
    Race: White - White/Caucasian/European Heritage | 5 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Any Non-serious Adverse Event (Non-SAE), Serious AE (SAE), Dose Limiting Toxicities (DLT), Dose Reductions or Delays and Withdrawals Due to Toxicities
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention or event associated with liver injury and impaired liver function were categorized as SAE. An event was considered a DLT if it occurred within the first 28 days of treatment, and met the DLT criteria unless it could be clearly established that the event was unrelated to treatment.
Time Frame: Up to 2 years
Population: All Treated Subjects Population: All participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Participants
  Non-SAEs | 5
  SAEs | 1
  DLT | 0
  Dose reductions or delays | 0
  Withdrawals due to toxicities | 0

2. Primary Outcome: Part 1: Change From Baseline in Platelets, Neutrophils, Monocytes, Lymphocytes, Leucocyte, Eosinophils and Basophils at Indicated Time-points
Description: Blood samples were collected from participants for evaluation of hematology parameters including platelets, neutrophils, monocytes, lymphocytes, leucocyte, eosinophils and basophils. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and Cycle 1(Days 1, 7, 15, 22), Cycle 2 (Days 1, 7, 15 ,22), Cycle 3 (Day 1), Cycle 4 (Day 1), Cycle 5 (Day 1) (each cycle of 28 days)
Population: All Treated Subjects Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
10^9 cells per liter
  Platelets, Cycle 1, Day 1, n=5 | -13.826 (16.2868)
  Platelets, Cycle 1, Day 7, n=5 | -17.984 (15.7398)
  Platelets, Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Platelets, Cycle 1, Day 15, n=4 | -19.250 (8.2614)
  Platelets, Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Platelets, Cycle 1, Day 22, n=3 | -20.667 (14.3643)
  Platelets, Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Platelets, Cycle 2, Day 1, n=3 | -16.000 (18.7350)
  Platelets, Cycle 2, Day 7, n=3: number analyzed (Participants) | 3
  Platelets, Cycle 2, Day 7, n=3 | -21.333 (28.3784)
  Platelets, Cycle 2, Day 15, n=3: number analyzed (Participants) | 3
  Platelets, Cycle 2, Day 15, n=3 | -24.333 (15.3731)
  Platelets, Cycle 2, Day 22, n=3: number analyzed (Participants) | 3
  Platelets, Cycle 2, Day 22, n=3 | -24.667 (19.3477)
  Platelets, Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Platelets, Cycle 3, Day 1, n=3 | -17.000 (14.1067)
  Platelets, Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Platelets, Cycle 4, Day 1, n=2 | -13.000 (4.2426)
  Platelets, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Platelets, Cycle 5, Day 1, n=1 | -11.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Neutrophils, Cycle 1, Day 1, n=5 | -0.019 (0.1298)
  Neutrophils, Cycle 1, Day 7, n=5 | 0.035 (0.2058)
  Neutrophils, Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Neutrophils, Cycle 1, Day 15, n=4 | 0.060 (0.3282)
  Neutrophils, Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Neutrophils, Cycle 1, Day 22, n=3 | 0.100 (0.1732)
  Neutrophils, Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Neutrophils, Cycle 2, Day 1, n=3 | 0.200 (0.3000)
  Neutrophils, Cycle 2, Day 7, n=3: number analyzed (Participants) | 3
  Neutrophils, Cycle 2, Day 7, n=3 | 0.300 (0.3606)
  Neutrophils, Cycle 2, Day 15, n=3: number analyzed (Participants) | 3
  Neutrophils, Cycle 2, Day 15, n=3 | 0.333 (0.3055)
  Neutrophils, Cycle 2, Day 22, n=3: number analyzed (Participants) | 3
  Neutrophils, Cycle 2, Day 22, n=3 | 0.267 (0.4041)
  Neutrophils, Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Neutrophils, Cycle 3, Day 1, n=3 | 0.267 (0.3215)
  Neutrophils, Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Neutrophils, Cycle 4, Day 1, n=2 | 0.650 (0.2121)
  Neutrophils, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Neutrophils, Cycle 5, Day 1, n=1 | 0.800 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Monocytes, Cycle 1, Day 1, n=5 | 0.017 (0.1359)
  Monocytes, Cycle 1, Day 7, n=5 | 0.059 (0.0853)
  Monocytes, Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Monocytes, Cycle 1, Day 15, n=4 | 0.100 (0.0816)
  Monocytes, Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Monocytes, Cycle 1, Day 22, n=3 | 12.633 (21.7086)
  Monocytes, Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Monocytes, Cycle 2, Day 1, n=3 | 0.267 (0.2517)
  Monocytes, Cycle 2, Day 7, n=3: number analyzed (Participants) | 3
  Monocytes, Cycle 2, Day 7, n=3 | 0.400 (0.6083)
  Monocytes, Cycle 2, Day 15, n=3: number analyzed (Participants) | 3
  Monocytes, Cycle 2, Day 15, n=3 | 0.633 (0.7095)
  Monocytes, Cycle 2, Day 22, n=3: number analyzed (Participants) | 3
  Monocytes, Cycle 2, Day 22, n=3 | 0.267 (0.2517)
  Monocytes, Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Monocytes, Cycle 3, Day 1, n=3 | 0.300 (0.1732)
  Monocytes, Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Monocytes, Cycle 4, Day 1, n=2 | 1.000 (0.1414)
  Monocytes, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Monocytes, Cycle 5, Day 1, n=1 | 1.600 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Lymphocytes, Cycle 1, Day 1, n=5 | -0.036 (0.0924)
  Lymphocytes, Cycle 1, Day 7, n=5 | 0.008 (0.1761)
  Lymphocytes, Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Lymphocytes, Cycle 1, Day 15, n=4 | -0.073 (0.0486)
  Lymphocytes, Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Lymphocytes, Cycle 1, Day 22, n=3 | -0.033 (0.0577)
  Lymphocytes, Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Lymphocytes, Cycle 2, Day 1, n=3 | -0.067 (0.1528)
  Lymphocytes, Cycle 2, Day 7, n=3: number analyzed (Participants) | 3
  Lymphocytes, Cycle 2, Day 7, n=3 | -0.033 (0.3055)
  Lymphocytes, Cycle 2, Day 15, n=3: number analyzed (Participants) | 3
  Lymphocytes, Cycle 2, Day 15, n=3 | 0.033 (0.3786)
  Lymphocytes, Cycle 2, Day 22, n=3: number analyzed (Participants) | 3
  Lymphocytes, Cycle 2, Day 22, n=3 | 0.033 (0.2082)
  Lymphocytes, Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Lymphocytes, Cycle 3, Day 1, n=3 | -0.067 (0.3055)
  Lymphocytes, Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Lymphocytes, Cycle 4, Day 1, n=2 | 0.200 (0.0000)
  Lymphocytes, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Lymphocytes, Cycle 5, Day 1, n=1 | 0.400 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Leucocytes, Cycle 1, Day 1, n=5 | -0.054 (0.1720)
  Leucocytes, Cycle 1, Day 7, n=5 | 0.154 (0.3257)
  Leucocytes, Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Leucocytes, Cycle 1, Day 15, n=4 | 0.032 (0.3208)
  Leucocytes, Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Leucocytes, Cycle 1, Day 22, n=3 | 0.267 (0.5132)
  Leucocytes, Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Leucocytes, Cycle 2, Day 1, n=3 | 0.433 (0.7234)
  Leucocytes, Cycle 2, Day 7, n=3: number analyzed (Participants) | 3
  Leucocytes, Cycle 2, Day 7, n=3 | 0.700 (1.3748)
  Leucocytes, Cycle 2, Day 15, n=3: number analyzed (Participants) | 3
  Leucocytes, Cycle 2, Day 15, n=3 | 1.033 (1.4572)
  Leucocytes, Cycle 2, Day 22, n=3: number analyzed (Participants) | 3
  Leucocytes, Cycle 2, Day 22, n=3 | 0.633 (0.9292)
  Leucocytes, Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Leucocytes, Cycle 3, Day 1, n=3 | 0.633 (0.9074)
  Leucocytes, Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Leucocytes, Cycle 4, Day 1, n=2 | 2.000 (0.0000)
  Leucocytes, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Leucocytes, Cycle 5, Day 1, n=1 | 2.900 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Eosinophils, Cycle 1, Day 1, n=5 | -0.000 (0.0009)
  Eosinophils, Cycle 1, Day 7, n=5 | 0.016 (0.0252)
  Eosinophils, Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Eosinophils, Cycle 1, Day 15, n=4 | -0.008 (0.0150)
  Eosinophils, Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Eosinophils, Cycle 1, Day 22, n=3 | 0.000 (0.0000)
  Eosinophils, Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Eosinophils, Cycle 2, Day 1, n=3 | 0.000 (0.0000)
  Eosinophils, Cycle 2, Day 7, n=3: number analyzed (Participants) | 3
  Eosinophils, Cycle 2, Day 7, n=3 | 0.000 (0.0000)
  Eosinophils, Cycle 2, Day 15, n=3: number analyzed (Participants) | 3
  Eosinophils, Cycle 2, Day 15, n=3 | 0.000 (0.0000)
  Eosinophils, Cycle 2, Day 22, n=3: number analyzed (Participants) | 3
  Eosinophils, Cycle 2, Day 22, n=3 | 0.000 (0.0000)
  Eosinophils, Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Eosinophils, Cycle 3, Day 1, n=3 | 0.000 (0.0000)
  Eosinophils, Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Eosinophils, Cycle 4, Day 1, n=2 | 0.050 (0.0707)
  Eosinophils, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Eosinophils, Cycle 5, Day 1, n=1 | 0.100 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Basophils, Cycle 1, Day 1, n=5 | 0.004 (0.0080)
  Basophils, Cycle 1, Day 7, n=5 | 0.017 (0.0323)
  Basophils, Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Basophils, Cycle 1, Day 15, n=4 | 0.003 (0.0050)
  Basophils, Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Basophils, Cycle 1, Day 22, n=3 | 0.000 (0.0000)
  Basophils, Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Basophils, Cycle 2, Day 1, n=3 | 0.000 (0.0000)
  Basophils, Cycle 2, Day 7, n=3: number analyzed (Participants) | 3
  Basophils, Cycle 2, Day 7, n=3 | 0.000 (0.0000)
  Basophils, Cycle 2, Day 15, n=3: number analyzed (Participants) | 3
  Basophils, Cycle 2, Day 15, n=3 | 0.000 (0.0000)
  Basophils, Cycle 2, Day 22, n=3: number analyzed (Participants) | 3
  Basophils, Cycle 2, Day 22, n=3 | 0.000 (0.0000)
  Basophils, Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Basophils, Cycle 3, Day 1, n=3 | 0.000 (0.0000)
  Basophils, Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Basophils, Cycle 4, Day 1, n=2 | 0.050 (0.0707)
  Basophils, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Basophils, Cycle 5, Day 1, n=1 | 0.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

3. Primary Outcome: Part 1: Change From Baseline in Mean Corpuscular Volume (MCV) at Indicated Time-points
Description: Blood samples were collected from participants for evaluation of hematology parameters including MCV. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Femtoliter
  Cycle 1, Day 1, n=5 | -0.280 (1.5450)
  Cycle 1, Day 7, n=4: number analyzed (Participants) | 4
  Cycle 1, Day 7, n=4 | -0.400 (1.9442)
  Cycle 1, Day 15, n=3: number analyzed (Participants) | 3
  Cycle 1, Day 15, n=3 | -0.267 (3.6679)
  Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Cycle 1, Day 22, n=3 | 0.400 (5.1730)
  Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 1, n=3 | 1.667 (6.0003)
  Cycle 2, Day 7, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 7, n=3 | 3.500 (6.3592)
  Cycle 2, Day 15, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 15, n=3 | 2.933 (7.3528)
  Cycle 2, Day 22, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 22, n=3 | 2.900 (9.0000)
  Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 3, Day 1, n=3 | 2.700 (9.7370)
  Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Cycle 4, Day 1, n=2 | 6.750 (6.2933)
  Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Cycle 5, Day 1, n=1 | 8.500 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

4. Primary Outcome: Part 1: Change From Baseline in Mean Corpuscular Hemoglobin (MCH) at Indicated Time-points
Description: Blood samples were collected from participants for evaluation of hematology parameters including MCH. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Picogram
  Cycle 1, Day 1, n=5 | -1.100 (2.8679)
  Cycle 1, Day 7, n=4: number analyzed (Participants) | 4
  Cycle 1, Day 7, n=4 | -1.350 (3.3000)
  Cycle 1, Day 15, n=3: number analyzed (Participants) | 3
  Cycle 1, Day 15, n=3 | -0.100 (1.1358)
  Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Cycle 1, Day 22, n=3 | 0.067 (1.5308)
  Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 1, n=3 | 0.833 (1.5177)
  Cycle 2, Day 7, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 7, n=3 | 1.067 (1.3796)
  Cycle 2, Day 15, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 15, n=3 | 0.900 (1.9672)
  Cycle 2, Day 22, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 22, n=3 | 0.767 (2.3798)
  Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 3, Day 1, n=3 | 0.933 (3.0665)
  Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Cycle 4, Day 1, n=2 | 1.950 (1.3435)
  Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Cycle 5, Day 1, n=1 | 2.200 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

5. Primary Outcome: Part 1: Change From Baseline in Mean Corpuscular Hemoglobin Concentration (MCHC) and Hemoglobin (Hb) at Indicated Time-points
Description: Blood samples were collected from participants for evaluation of hematology parameters including MCHC and Hb. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Grams per liter
  MCHC, Cycle 1, Day 1, n=5 | -10.400 (29.3053)
  MCHC, Cycle 1, Day 7, n=4: number analyzed (Participants) | 4
  MCHC, Cycle 1, Day 7, n=4 | -12.500 (35.8190)
  MCHC, Cycle 1, Day 15, n=3: number analyzed (Participants) | 3
  MCHC, Cycle 1, Day 15, n=3 | 0.333 (2.0817)
  MCHC, Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  MCHC, Cycle 1, Day 22, n=3 | 0.000 (8.1854)
  MCHC, Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  MCHC, Cycle 2, Day 1, n=3 | 3.667 (6.6583)
  MCHC, Cycle 2, Day 7, n=3: number analyzed (Participants) | 3
  MCHC, Cycle 2, Day 7, n=3 | -1.000 (12.4900)
  MCHC, Cycle 2, Day 15, n=3: number analyzed (Participants) | 3
  MCHC, Cycle 2, Day 15, n=3 | 0.000 (7.8102)
  MCHC, Cycle 2, Day 22, n=3: number analyzed (Participants) | 3
  MCHC, Cycle 2, Day 22, n=3 | -2.000 (8.6603)
  MCHC, Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  MCHC, Cycle 3, Day 1, n=3 | 1.333 (6.0277)
  MCHC, Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  MCHC, Cycle 4, Day 1, n=2 | -3.500 (9.1924)
  MCHC, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  MCHC, Cycle 5, Day 1, n=1 | -8.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Hb, Cycle 1, Day 1, n=5 | -2.000 (7.0000)
  Hb, Cycle 1, Day 7, n=5 | -4.200 (11.3666)
  Hb, Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Hb, Cycle 1, Day 15, n=4 | -5.000 (11.8040)
  Hb, Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Hb, Cycle 1, Day 22, n=3 | 2.000 (2.6458)
  Hb, Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Hb, Cycle 2, Day 1, n=3 | -3.667 (12.5831)
  Hb, Cycle 2, Day 7, n=3: number analyzed (Participants) | 3
  Hb, Cycle 2, Day 7, n=3 | 2.000 (13.4536)
  Hb, Cycle 2, Day 15, n=3: number analyzed (Participants) | 3
  Hb, Cycle 2, Day 15, n=3 | 0.333 (16.5630)
  Hb, Cycle 2, Day 22, n=3: number analyzed (Participants) | 3
  Hb, Cycle 2, Day 22, n=3 | -3.000 (5.2915)
  Hb, Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Hb, Cycle 3, Day 1, n=3 | -2.333 (7.2342)
  Hb, Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Hb, Cycle 4, Day 1, n=2 | 7.000 (4.2426)
  Hb, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Hb, Cycle 5, Day 1, n=1 | 6.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

6. Primary Outcome: Part 1: Change From Baseline in Hematocrit at Indicated Time-points
Description: Blood samples were collected from participants for evaluation of hematology parameters including Hematocrit. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Proportion of red blood cells in blood
  Cycle 1, Day 1, n=5 | 0.001 (0.0334)
  Cycle 1, Day 7, n=5 | -0.008 (0.0525)
  Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Cycle 1, Day 15, n=4 | -0.018 (0.0401)
  Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Cycle 1, Day 22, n=3 | 0.007 (0.0100)
  Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 1, n=3 | -0.014 (0.0396)
  Cycle 2, Day 7, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 7, n=3 | 0.007 (0.0448)
  Cycle 2, Day 15, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 15, n=3 | 0.002 (0.0520)
  Cycle 2, Day 22, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 22, n=3 | -0.009 (0.0206)
  Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 3, Day 1, n=3 | -0.008 (0.0244)
  Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Cycle 4, Day 1, n=2 | 0.024 (0.0191)
  Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Cycle 5, Day 1, n=1 | 0.023 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

7. Primary Outcome: Part 1: Change From Baseline in Erythrocytes at Indicated Time-points
Description: Blood samples were collected from participants for evaluation of hematology parameters including erythrocytes. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^12 cells per Liter
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
10^12 cells per Liter
  Cycle 1, Day 1, n=5 | 0.030 (0.3489)
  Cycle 1, Day 7, n=5 | -0.058 (0.5363)
  Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Cycle 1, Day 15, n=4 | -0.138 (0.3216)
  Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Cycle 1, Day 22, n=3 | 0.077 (0.0643)
  Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 1, n=3 | -0.193 (0.2558)
  Cycle 2, Day 7, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 7, n=3 | -0.017 (0.2996)
  Cycle 2, Day 15, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 15, n=3 | -0.063 (0.3402)
  Cycle 2, Day 22, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 22, n=3 | -0.173 (0.1901)
  Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 3, Day 1, n=3 | -0.160 (0.2425)
  Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Cycle 4, Day 1, n=2 | 0.060 (0.0141)
  Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Cycle 5, Day 1, n=1 | 0.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

8. Primary Outcome: Part 1: Change From Baseline in Percent Reticulocytes at Indicated Time-points
Description: Blood samples were collected from participants for evaluation of hematology parameters including percent reticulocytes. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and Cycle 1(Days 1, 7, 15, 22), Cycle 2 (Days 1, 7, 15 ,22), Cycle 3 (Day 1), Cycle 4 (Day 1) (each cycle of 28 days)
Population: All Treated Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 1
Percentage of reticulocytes
  Cycle 1, Day 7 | 0.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Cycle 1, Day 22 | -0.100 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Cycle 2, Day 1 | -0.100 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Cycle 2, Day 7 | 0.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Cycle 2, Day 15 | 0.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Cycle 3, Day 1 | -0.100 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Cycle 4, Day 1 | -0.100 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

9. Primary Outcome: Part 1: Change From Baseline in Blast/Leukocytes at Indicated Time-points
Description: Blood samples were collected from participants for evaluation of hematology parameters including blast/leukocytes. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and Day 1 of Cycle 1 (Cycle of 28 days)
Population: All Treated Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio of blasts to leukocytes
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 1
Ratio of blasts to leukocytes | 0.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

10. Primary Outcome: Part 1: Change From Baseline in Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Lactate Dehydrogenase (LDH) and Gamma Glutamyl Transferase (GGT) at Indicated Time-points
Description: Blood samples were collected from participants for evaluation of clinical chemistry parameters including ALT, ALP, AST, LDH and GGT. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
International unit per liter (IU/L)
  ALT, Cycle 1, Day 1, n=4: number analyzed (Participants) | 4
  ALT, Cycle 1, Day 1, n=4 | -10.000 (18.1292)
  ALT Cycle 1, Day 7, n=5 | -3.000 (13.5093)
  ALT Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  ALT Cycle 1, Day 15, n=4 | -6.250 (15.5000)
  ALT Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  ALT Cycle 1, Day 22, n=3 | 1.333 (15.1767)
  ALT Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  ALT Cycle 2, Day 1, n=3 | 3.000 (39.5095)
  ALT Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  ALT Cycle 3, Day 1, n=3 | 3.333 (42.0040)
  ALT Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  ALT Cycle 4, Day 1, n=2 | 33.000 (1.4142)
  ALT Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  ALT Cycle 5, Day 1, n=1 | 3.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  ALP, Cycle 1, Day 1, n=4: number analyzed (Participants) | 4
  ALP, Cycle 1, Day 1, n=4 | -4.750 (3.2016)
  ALP Cycle 1, Day 7, n=5 | -6.800 (10.3053)
  ALP Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  ALP Cycle 1, Day 15, n=4 | -4.250 (22.3961)
  ALP Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  ALP Cycle 1, Day 22, n=3 | 8.000 (21.6564)
  ALP Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  ALP Cycle 2, Day 1, n=3 | 23.667 (62.5007)
  ALP Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  ALP Cycle 3, Day 1, n=3 | 15.667 (31.3422)
  ALP Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  ALP Cycle 4, Day 1, n=2 | 18.500 (60.1041)
  ALP Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  ALP Cycle 5, Day 1, n=1 | 21.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  AST, Cycle 1, Day 1, n=4: number analyzed (Participants) | 4
  AST, Cycle 1, Day 1, n=4 | -6.750 (14.8633)
  AST Cycle 1, Day 7, n=5 | -3.200 (9.3381)
  AST Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  AST Cycle 1, Day 15, n=4 | -3.250 (17.6517)
  AST Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  AST Cycle 1, Day 22, n=3 | 3.000 (27.5136)
  AST Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  AST Cycle 2, Day 1, n=3 | -0.333 (30.9246)
  AST Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  AST Cycle 3, Day 1, n=3 | -3.667 (38.5530)
  AST Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  AST Cycle 4, Day 1, n=2 | 22.000 (21.2132)
  AST Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  AST Cycle 5, Day 1, n=1 | 16.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  LDH, Cycle 1, Day 1, n=4: number analyzed (Participants) | 4
  LDH, Cycle 1, Day 1, n=4 | 4.000 (90.9395)
  LDH Cycle 1, Day 7, n=5 | -31.200 (47.2515)
  LDH Cycle 1, Day 15, n=3: number analyzed (Participants) | 3
  LDH Cycle 1, Day 15, n=3 | 4.000 (22.6053)
  LDH Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  LDH Cycle 1, Day 22, n=3 | -12.000 (47.5710)
  LDH Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  LDH Cycle 2, Day 1, n=3 | -18.333 (55.4106)
  LDH Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  LDH Cycle 3, Day 1, n=3 | -20.667 (62.7402)
  LDH Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  LDH Cycle 4, Day 1, n=2 | 12.500 (3.5355)
  LDH Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  LDH Cycle 5, Day 1, n=1 | 11.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  GGT, Cycle 1, Day 1, n=1: number analyzed (Participants) | 1
  GGT, Cycle 1, Day 1, n=1 | -17.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  GGT Cycle 1, Day 7, n=2: number analyzed (Participants) | 2
  GGT Cycle 1, Day 7, n=2 | -7.500 (9.1924)
  GGT Cycle 1, Day 22, n=1: number analyzed (Participants) | 1
  GGT Cycle 1, Day 22, n=1 | 0.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  GGT Cycle 2, Day 1, n=1: number analyzed (Participants) | 1
  GGT Cycle 2, Day 1, n=1 | 3.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  GGT Cycle 3, Day 1, n=1: number analyzed (Participants) | 1
  GGT Cycle 3, Day 1, n=1 | 8.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  GGT Cycle 4, Day 1, n=1: number analyzed (Participants) | 1
  GGT Cycle 4, Day 1, n=1 | 5.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

11. Primary Outcome: Part 1: Change From Baseline in Calcium, Chloride, Glucose, Potassium, Sodium, Phosphate and Urea Nitrogen at Indicated Time-points
Description: Blood samples were collected from participants for evaluation of clinical chemistry parameters including calcium, chloride, glucose, potassium, sodium, phosphate and urea nitrogen. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Millimoles per liter (mmol/L)
  Calcium, Cycle 1, Day 1, n=3: number analyzed (Participants) | 3
  Calcium, Cycle 1, Day 1, n=3 | -0.008 (0.0520)
  Calcium Cycle 1, Day 7, n=4: number analyzed (Participants) | 4
  Calcium Cycle 1, Day 7, n=4 | -0.075 (0.0535)
  Calcium Cycle 1, Day 15, n=3: number analyzed (Participants) | 3
  Calcium Cycle 1, Day 15, n=3 | -0.066 (0.0758)
  Calcium Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Calcium Cycle 1, Day 22, n=3 | -0.033 (0.0624)
  Calcium Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Calcium Cycle 2, Day 1, n=3 | -0.067 (0.0144)
  Calcium Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Calcium Cycle 3, Day 1, n=3 | -0.183 (0.1523)
  Calcium Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Calcium Cycle 4, Day 1, n=2 | -0.050 (0.0700)
  Calcium, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Calcium, Cycle 5, Day 1, n=1 | -0.050 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Chloride, Cycle 1, Day 1, n=4: number analyzed (Participants) | 4
  Chloride, Cycle 1, Day 1, n=4 | -0.750 (0.5000)
  Chloride Cycle 1, Day 7, n=5 | 0.600 (4.3932)
  Chloride Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Chloride Cycle 1, Day 15, n=4 | 0.250 (2.5000)
  Chloride Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Chloride Cycle 1, Day 22, n=3 | 0.333 (1.1547)
  Chloride Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Chloride Cycle 2, Day 1, n=3 | 0.333 (1.5275)
  Chloride Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Chloride Cycle 3, Day 1, n=3 | -0.333 (1.5275)
  Chloride Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Chloride Cycle 4, Day 1, n=2 | 0.000 (2.8284)
  Chloride, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Chloride, Cycle 5, Day 1, n=1 | 0.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Glucose, Cycle 1, Day 1, n=4: number analyzed (Participants) | 4
  Glucose, Cycle 1, Day 1, n=4 | 0.527 (1.9147)
  Glucose Cycle 1, Day 7, n=5 | -0.333 (1.5357)
  Glucose Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Glucose Cycle 1, Day 15, n=4 | 0.014 (0.7971)
  Glucose Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Glucose Cycle 1, Day 22, n=3 | 0.870 (0.9309)
  Glucose Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Glucose Cycle 2, Day 1, n=3 | 1.924 (2.1037)
  Glucose Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Glucose Cycle 3, Day 1, n=3 | 1.628 (2.8543)
  Glucose Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Glucose Cycle 4, Day 1, n=2 | 1.027 (1.2954)
  Glucose, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Glucose, Cycle 5, Day 1, n=1 | 1.110 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Potassium, Cycle 1, Day 1, n=4: number analyzed (Participants) | 4
  Potassium, Cycle 1, Day 1, n=4 | 0.325 (0.5315)
  Potassium Cycle 1, Day 7, n=5 | 0.000 (0.4528)
  Potassium Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Potassium Cycle 1, Day 15, n=4 | -0.025 (0.4272)
  Potassium Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Potassium Cycle 1, Day 22, n=3 | 0.067 (0.2887)
  Potassium Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Potassium Cycle 2, Day 1, n=3 | 0.067 (0.1528)
  Potassium Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Potassium Cycle 3, Day 1, n=3 | -0.367 (0.3786)
  Potassium Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Potassium Cycle 4, Day 1, n=2 | 0.050 (0.0707)
  Potassium, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Potassium, Cycle 5, Day 1, n=1 | 0.500 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Sodium, Cycle 1, Day 1, n=4: number analyzed (Participants) | 4
  Sodium, Cycle 1, Day 1, n=4 | -1.750 (1.2583)
  Sodium Cycle 1, Day 7, n=5 | -1.000 (2.2361)
  Sodium Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Sodium Cycle 1, Day 15, n=4 | -2.000 (2.4495)
  Sodium Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Sodium Cycle 1, Day 22, n=3 | -0.667 (2.0817)
  Sodium Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Sodium Cycle 2, Day 1, n=3 | 0.333 (0.5774)
  Sodium Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Sodium Cycle 3, Day 1, n=3 | -1.000 (5.0000)
  Sodium Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Sodium Cycle 4, Day 1, n=2 | -0.500 (2.1213)
  Sodium, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Sodium, Cycle 5, Day 1, n=1 | 0.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Urea nitrogen, Cycle 1, Day 1, n=3: number analyzed (Participants) | 3
  Urea nitrogen, Cycle 1, Day 1, n=3 | 2.701 (2.3181)
  Urea nitrogen Cycle 1, Day 7, n=4: number analyzed (Participants) | 4
  Urea nitrogen Cycle 1, Day 7, n=4 | 1.214 (3.4779)
  Urea nitrogen Cycle 1, Day 15, n=3: number analyzed (Participants) | 3
  Urea nitrogen Cycle 1, Day 15, n=3 | 1.547 (3.3171)
  Urea nitrogen Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Urea nitrogen Cycle 1, Day 22, n=3 | 1.309 (3.8173)
  Urea nitrogen Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Urea nitrogen Cycle 2, Day 1, n=3 | 0.238 (2.1519)
  Urea nitrogen Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Urea nitrogen Cycle 3, Day 1, n=3 | -1.190 (1.7610)
  Urea nitrogen Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Urea nitrogen Cycle 4, Day 1, n=2 | -0.535 (1.2622)
  Urea nitrogen, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Urea nitrogen, Cycle 5, Day 1, n=1 | -1.428 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Phosphate, Cycle 1, Day 1, n=1: number analyzed (Participants) | 1
  Phosphate, Cycle 1, Day 1, n=1 | 0.194 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Phosphate Cycle 1, Day 7, n=2: number analyzed (Participants) | 2
  Phosphate Cycle 1, Day 7, n=2 | -0.081 (0.1598)
  Phosphate Cycle 1, Day 22, n=1: number analyzed (Participants) | 1
  Phosphate Cycle 1, Day 22, n=1 | -0.032 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Phosphate Cycle 2, Day 1, n=1: number analyzed (Participants) | 1
  Phosphate Cycle 2, Day 1, n=1 | 0.194 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Phosphate Cycle 3, Day 1, n=1: number analyzed (Participants) | 1
  Phosphate Cycle 3, Day 1, n=1 | 0.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Phosphate Cycle 4, Day 1, n=1: number analyzed (Participants) | 1
  Phosphate Cycle 4, Day 1, n=1 | 0.032 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

12. Primary Outcome: Part 1: Change From Baseline in Albumin and Protein at Indicated Time Points
Description: Blood samples were collected from participants for evaluation of clinical chemistry parameters including Albumin and Protein. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
G/L
  Albumin, Cycle 1, Day 1, n=4: number analyzed (Participants) | 4
  Albumin, Cycle 1, Day 1, n=4 | -1.250 (2.2174)
  Albumin Cycle 1, Day 7, n=4: number analyzed (Participants) | 4
  Albumin Cycle 1, Day 7, n=4 | -1.250 (2.5000)
  Albumin Cycle 1, Day 15, n=3: number analyzed (Participants) | 3
  Albumin Cycle 1, Day 15, n=3 | -1.667 (1.5275)
  Albumin Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Albumin Cycle 1, Day 22, n=3 | -1.333 (0.5774)
  Albumin Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Albumin Cycle 2, Day 1, n=3 | -1.667 (2.0817)
  Albumin Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Albumin Cycle 3, Day 1, n=3 | -6.000 (6.2450)
  Albumin Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Albumin Cycle 4, Day 1, n=2 | 0.000 (1.4142)
  Albumin Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Albumin Cycle 5, Day 1, n=1 | 1.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants
  Protein, Cycle 1, Day 1, n=4: number analyzed (Participants) | 4
  Protein, Cycle 1, Day 1, n=4 | -3.250 (3.8622)
  Protein Cycle 1, Day 7, n=5 | -3.200 (4.3243)
  Protein Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Protein Cycle 1, Day 15, n=4 | -1.500 (4.4347)
  Protein Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Protein Cycle 1, Day 22, n=3 | -1.667 (1.1547)
  Protein Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Protein Cycle 2, Day 1, n=3 | -3.333 (5.8595)
  Protein Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Protein Cycle 3, Day 1, n=3 | -7.333 (6.8069)
  Protein Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Protein Cycle 4, Day 1, n=2 | -2.000 (2.8284)
  Protein Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Protein Cycle 5, Day 1, n=1 | 0.000 (NA) — Standard deviation could not be calculated due to insufficient number of participants

13. Primary Outcome: Part 1: Change From Baseline in Partial Pressure Carbon Dioxide (pCO2) at Indicated Time Points
Description: Blood samples were collected from participants for evaluation of clinical chemistry parameters including pCO2. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and Day 1 of Cycle 1 (cycle of 28 days)
Population: All Treated Subjects Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilopascal
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 1
Kilopascal | 0.173 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

14. Primary Outcome: Part 1: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Indicated Time-points
Description: Vital signs including SBP and DBP were measured after resting for at least 5 minutes in a semi-supine position. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and Cycle 1 (Days 7, 15), Cycle 2 (Day 1), Cycle 3 (Day 1), Cycle 4 (Day 1), Cycle 5 (Day 1) (each cycle of 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Millimeters of mercury
  SBP, Cycle 1, Day 7, n=5 | -10.2 (4.76)
  SBP, Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  SBP, Cycle 1, Day 15, n=4 | -13.5 (3.87)
  SBP, Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  SBP, Cycle 2, Day 1, n=3 | -4.7 (3.79)
  SBP, Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  SBP, Cycle 3, Day 1, n=3 | -3.7 (8.39)
  SBP, Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  SBP, Cycle 4, Day 1, n=2 | -5.0 (2.83)
  SBP, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  SBP, Cycle 5, Day 1, n=1 | -6.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  DBP, Cycle 1, Day 7, n=5 | -2.6 (8.62)
  DBP, Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  DBP, Cycle 1, Day 15, n=4 | -3.5 (4.04)
  DBP, Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  DBP, Cycle 2, Day 1, n=3 | -7.3 (10.02)
  DBP, Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  DBP, Cycle 3, Day 1, n=3 | 2.7 (4.73)
  DBP, Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  DBP, Cycle 4, Day 1, n=2 | 3.0 (7.07)
  DBP, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  DBP, Cycle 5, Day 1, n=1 | -4.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

15. Primary Outcome: Part 1: Change From Baseline in Heart Rate at Indicated Time-points
Description: Vital signs including heart rate was measured after resting for at least 5 minutes in a semi-supine position. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: as for outcome 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Beats per minute
  Cycle 1, Day 7, n=5 | 4.8 (6.69)
  Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Cycle 1, Day 15, n=4 | -2.5 (7.42)
  Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 1, n=3 | -6.3 (2.89)
  Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 3, Day 1, n=3 | -1.0 (9.00)
  Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Cycle 4, Day 1, n=2 | -2.0 (8.49)
  Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Cycle 5, Day 1, n=1 | -1.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

16. Primary Outcome: Part 1: Change From Baseline in Respiratory Rate at Indicated Time-points
Description: Vital signs including respiratory rate was measured after resting for at least 5 minutes in a semi-supine position. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: as for outcome 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Breaths per minute
  Cycle 1, Day 7, n=5 | -0.4 (1.14)
  Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Cycle 1, Day 15, n=4 | -0.5 (1.00)
  Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 1, n=3 | -1.0 (1.00)
  Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 3, Day 1, n=3 | -0.3 (1.53)
  Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Cycle 4, Day 1, n=2 | -0.5 (0.71)
  Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Cycle 5, Day 1, n=1 | -1.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

17. Primary Outcome: Part 1: Change From Baseline in Body Temperature at Indicated Time-points
Description: Vital signs including body temperature was measured after resting for at least 5 minutes in a semi-supine position. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: as for outcome 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Celsius
  Cycle 1, Day 7, n=5 | 0.14 (0.279)
  Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Cycle 1, Day 15, n=4 | 0.10 (0.216)
  Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 1, n=3 | 0.27 (0.231)
  Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 3, Day 1, n=3 | 0.20 (0.300)
  Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Cycle 4, Day 1, n=2 | 0.10 (0.283)
  Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Cycle 5, Day 1, n=1 | -0.20 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

18. Primary Outcome: Part 1: Change From Baseline in Electrocardiogram (ECG) Mean Heart Rate at Indicated Time-points
Description: Single 12-lead ECG was obtained at designated time points during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT (QTc) intervals. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and Cycle 1 (Days 1, 7), Cycle 2 (Day 1), Cycle 3 (Day 1), Cycle 4 (Day 1), Cycle 5 (Day 1) (each cycle of 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Beats per minute
  Cycle 1, Day 1, n=2: number analyzed (Participants) | 2
  Cycle 1, Day 1, n=2 | 2.0 (2.83)
  Cycle 1, Day 7, n=5 | -1.0 (11.94)
  Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 1, n=3 | -5.3 (5.51)
  Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Cycle 3, Day 1, n=3 | 2.3 (10.02)
  Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Cycle 4, Day 1, n=2 | -3.0 (9.90)
  Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Cycle 5, Day 1, n=1 | -7.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

19. Primary Outcome: Part 1: Change From Baseline in ECG PR Interval, QRS Duration, QT Interval, QTc Corrected by Bazett's Formula (QTcB) and QTc Corrected by Fridericia's Formula (QTcF) at Indicated Time-points
Description: Single 12-lead ECG was obtained at designated time points during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and Cycle 1 (Days 1,7), Cycle 2 (Day 1), Cycle 3 (Day 1), Cycle 4 (Day 1), Cycle 5 (Day 1) (each cycle of 28 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Milliseconds
  PR interval, Cycle 1, Day 1, n=2: number analyzed (Participants) | 2
  PR interval, Cycle 1, Day 1, n=2 | 0.0 (0.00)
  PR interval, Cycle 1, Day 7, n=5 | 39.8 (88.34)
  PR interval, Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  PR interval, Cycle 2, Day 1, n=3 | 6.0 (9.17)
  PR interval, Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  PR interval, Cycle 3, Day 1, n=3 | 0.7 (8.08)
  PR interval, Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  PR interval, Cycle 4, Day 1, n=2 | 6.0 (14.14)
  PR interval, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  PR interval, Cycle 5, Day 1, n=1 | 12.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  QRS duration, Cycle 1, Day 1, n=2: number analyzed (Participants) | 2
  QRS duration, Cycle 1, Day 1, n=2 | -1.0 (4.24)
  QRS duration, Cycle 1, Day 7, n=5 | -17.2 (39.61)
  QRS duration, Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  QRS duration, Cycle 2, Day 1, n=3 | 2.0 (2.00)
  QRS duration, Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  QRS duration, Cycle 3, Day 1, n=3 | 3.3 (1.15)
  QRS duration, Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  QRS duration, Cycle 4, Day 1, n=2 | -1.0 (1.41)
  QRS duration, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  QRS duration, Cycle 5, Day 1, n=1 | -8.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  QT interval, Cycle 1, Day 1, n=2: number analyzed (Participants) | 2
  QT interval, Cycle 1, Day 1, n=2 | 0.0 (0.00)
  QT interval, Cycle 1, Day 7, n=5 | -5.6 (29.37)
  QT interval, Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  QT interval, Cycle 2, Day 1, n=3 | 24.7 (18.58)
  QT interval, Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  QT interval, Cycle 3, Day 1, n=3 | 2.0 (18.00)
  QT interval, Cycle 4, Day 1, n=1: number analyzed (Participants) | 1
  QT interval, Cycle 4, Day 1, n=1 | -4.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  QT interval, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  QT interval, Cycle 5, Day 1, n=1 | 14.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  QTcB interval, Cycle 1, Day 1, n=2: number analyzed (Participants) | 2
  QTcB interval, Cycle 1, Day 1, n=2 | 7.0 (9.90)
  QTcB interval, Cycle 1, Day 7, n=2: number analyzed (Participants) | 2
  QTcB interval, Cycle 1, Day 7, n=2 | -35.5 (82.73)
  QTcF interval, Cycle 1, Day 1, n=2: number analyzed (Participants) | 2
  QTcF interval, Cycle 1, Day 1, n=2 | 4.5 (6.36)
  QTcF interval, Cycle 1, Day 7, n=5 | -9.4 (38.12)
  QTcF interval, Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  QTcF interval, Cycle 2, Day 1, n=3 | 8.0 (5.57)
  QTcF interval, Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  QTcF interval, Cycle 3, Day 1, n=3 | 13.0 (18.52)
  QTcF interval, Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  QTcF interval, Cycle 4, Day 1, n=2 | -6.0 (19.80)
  QTcF interval, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  QTcF interval, Cycle 5, Day 1, n=1 | -8.0 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

20. Primary Outcome: Part 1: Number of Participants With Abnormal Findings During Physical Examination
Description: A complete physical examination included, at a minimum, assessment of the Cardiovascular, Respiratory, Gastrointestinal and Neurological systems. A brief physical examination included, at a minimum assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen). This analysis was planned but data was not captured in the database. Abnormal changes were captured as adverse events if they were clinically significant.
Time Frame: Up to 2 years
Population: All Treated Subjects Population. This analysis was planned but data was not captured in the database.
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 0

21. Primary Outcome: Part 2: Percentage of Participants With Investigator-assessed Best Response Assessed by Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants achieving a confirmed Complete Remission (CR) or Partial Remission (PR) or Marrow Complete Remission (mCR) or confirmed Hematologic Improvement (HI) or Stable Disease (SD) prior to new anti-cancer therapy and crossover on the All Treated Subjects Population. Participants with Not Evaluable or missing response were to be treated as non-responders. International Working Group (IWG) criteria, 2006 was to be used to evaluate response.
Time Frame: Up to 2.5 years
Population: All Treated Subjects Population. Data was not collected for this endpoint as study was terminated during Part 1 and Part 2 was not initiated.
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

22. Primary Outcome: Part 2: Percentage of Participants With Investigator-assessed Best Response Assessed by Objective Response Rate (ORR)
Description: Objective response rate was defined as the percentage of participants who achieved CR or PR or mCR or HI prior to new anti-cancer therapy on the All Treated Subjects Population. Participants with Not Evaluable or missing response were to be treated as non-responders. IWG criteria, 2006 was to be used to evaluate response.
Time Frame: Up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Part 1: Percentage of Participants With Investigator-assessed Best Response Assessed by Clinical Benefit Rate (CBR)
Description: Clinical Benefit Rate was defined as the percentage of participants achieving a confirmed Complete Remission (CR) or Partial Remission (PR) or Marrow Complete Remission (mCR) or confirmed Hematologic Improvement (HI) or Stable Disease (SD) prior to new anti-cancer therapy and crossover on the All Treated Subjects Population. Participants with Not Evaluable or missing response were treated as non-responders. International Working Group (IWG) criteria, 2006 was used to evaluate response.
Time Frame: Up to 2 years
Population: All Treated Subjects Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Percentage of Participants | 40 [5.3 to 85.3]

24. Secondary Outcome: Part 1: Percentage of Participants With Investigator-assessed Best Response Assessed by Objective Response Rate (ORR)
Description: Objective Response Rate was defined as the percentage of participants who achieved Complete Remission (CR) or Partial Remission (PR) or Marrow Complete Remission (mCR) or confirmed Hematologic Improvement (HI) prior to new anti-cancer therapy on the All Treated Subjects Population. Participants with Not Evaluable or missing response were treated as non-responders. International Working Group (IWG) criteria, 2006 was used to evaluate response.
Time Frame: Up to 2 years
Population: All Treated Subjects Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Percentage of Participants | 20 [0.5 to 71.6]

25. Secondary Outcome: Part 1: Plasma Concentration of GSK2879552
Description: Blood samples were collected at indicated time points to evaluate concentration of GSK2879552. Each Pharmacokinetic (PK) sample was collected as close as possible to the planned time relative to the dose (i.e., time zero) administered to the participant on PK days. PK Concentration Population consisted of all participants in the All Treated Subject Population for whom a blood sample for pharmacokinetics was obtained and analyzed.
Time Frame: Cycle 1, Day 1: pre-dose, 0.5, 1, 3 hour; pre-dose on Days 2,4; Day 7: pre-dose, 0.5, 1, 3 hour; Day 15: pre-dose, 0.5-1 hour post-dose; pre-dose on Day 22; Cycle 2: pre-dose on Days 1, 7, 15, 22; Pre-dose on Day 1 of Cycles 3,4,5 (each cycle of 28 days)
Population: PK Concentration Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Nanograms per milliliter
  Cycle 1, Day 1, pre-dose, n=5 | 0.00 (NA) — All concentration values were less than the lower limit of quantification, therefore they have been imputed with 0 because they were so small. Hence, standard deviation was not calculated as it would result to "0" and would be misleading.
  Cycle 1, Day 1, 0.5 hour, n=4: number analyzed (Participants) | 4
  Cycle 1, Day 1, 0.5 hour, n=4 | 11.79 (9.270)
  Cycle 1, Day 1, 1 hour, n=5 | 8.18 (4.830)
  Cycle 1, Day 1, 3 hour, n=5 | 6.40 (1.990)
  Cycle 1, Day 2, pre-dose, n=5 | 1.03 (0.409)
  Cycle 1, Day 4, pre-dose, n=5 | 1.87 (0.716)
  Cycle 1, Day 7, pre-dose, n=5 | 1.97 (0.553)
  Cycle 1, Day 7, 0.5 hour, n=5 | 9.58 (8.395)
  Cycle 1, Day 7, 1 hour, n=5 | 9.17 (4.4777)
  Cycle 1, Day 7, 3 hour, n=5 | 8.58 (3.595)
  Cycle 1, Day 15, pre-dose, n=3: number analyzed (Participants) | 3
  Cycle 1, Day 15, pre-dose, n=3 | 2.00 (0.798)
  Cycle 1, Day 15, 0.5-1 hour, n=3: number analyzed (Participants) | 3
  Cycle 1, Day 15, 0.5-1 hour, n=3 | 13.39 (0.798)
  Cycle 1, Day 22, pre-dose, n=3: number analyzed (Participants) | 3
  Cycle 1, Day 22, pre-dose, n=3 | 1.89 (0.723)
  Cycle 2, Day 1, pre-dose, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 1, pre-dose, n=3 | 2.16 (0.843)
  Cycle 2, Day 7, pre-dose, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 7, pre-dose, n=3 | 1.81 (0.585)
  Cycle 2, Day 15, pre-dose, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 15, pre-dose, n=3 | 2.33 (1.135)
  Cycle 2, Day 22, pre-dose, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 22, pre-dose, n=3 | 2.11 (0.709)
  Cycle 3, Day 1, pre-dose, n=3: number analyzed (Participants) | 3
  Cycle 3, Day 1, pre-dose, n=3 | 1.99 (0.802)
  Cycle 4, Day 1, pre-dose, n=2: number analyzed (Participants) | 2
  Cycle 4, Day 1, pre-dose, n=2 | 1.63 (0.085)
  Cycle 5, Day 1, pre-dose, n=1: number analyzed (Participants) | 1
  Cycle 5, Day 1, pre-dose, n=1 | 1.97 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

26. Secondary Outcome: Part 1: Plasma Concentration of Azacitidine
Description: Blood samples were to be collected at indicated time points to evaluate concentration of Azacitidine.
Time Frame: as for outcome 25
Population: PK Concentration Population. Data was not collected due to blood samples were not collected as participants were not enrolled in GSK2879552 + Azacitidine arm due to early termination of the study.
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 0

27. Secondary Outcome: Part 1: Duration of Response
Description: Duration of response is defined as the subset of participants (responders) who show a response (CR, mCR, PR, or HI), the time from first documented evidence of response until the first documented sign of disease progression or death. If no disease progression or death, the DOR was to be censored at last disease assessment.
Time Frame: Up to 2 years
Population: All Treated Subjects Population. Data was not collected for this endpoint as DOR could not be calculated because of the early termination of the study did not allow for this endpoint to be observed.
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 0

28. Secondary Outcome: Part 1: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the time from first treatment dose until the first documented sign of disease progression or death. If the participant missed more than one visit prior to the date of documented events, PFS was censored at the last adequate assessment prior to missing. Otherwise, if the participant did not have a documented date of events, PFS was censored at the date of the last adequate assessment.
Time Frame: Up to 2 years
Population: All Treated Subjects Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Weeks | 22.4 [4.3 to 22.4]

29. Secondary Outcome: Part 1: Overall Survival
Description: Overall survival (OS) is defined as the time from first treatment dose until death due to any reason. For the analysis of overall survival (OS), the last date of known contact was used for those participants who had not died at the time of analysis; such participants were considered censored.
Time Frame: Up to 2 years
Population: All Treated Subjects Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Weeks | 22.4 [16.4 to NA] — The data and very small number of participants did not allow meaningful calculation of the upper limit of 95% Confidence Interval.

30. Secondary Outcome: Part 1: Proportion of Participants With Disease Progression to Acute Myeloblastic Leukemia (AML)
Description: The proportion of participants with disease progression to AML is defined as the percentage of participants experiencing AML on the All Treated Subjects Population.
Time Frame: Up to 2 years
Population: All Treated Subjects Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Percentage of Participants | 40

31. Secondary Outcome: Part 1: Time to AML Progression
Description: Time to AML progression is defined as the time from first treatment dose until AML progression or crossover if using the All Treated Subjects Population. For the analysis of time to AML, if the participant did not experience AML, time to AML was censored at the last treatment prior to the initiation of anti-cancer therapy or crossover.
Time Frame: Up to 2 years
Population: All Treated Subjects Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Weeks | 22.4 [4.3 to 22.4]

32. Secondary Outcome: Part 1: Number of Participants With Documented Platelet and Red Blood Cell (RBC) Transfusions Per Month
Description: Number of participants with documented platelet and RBC transfusions have been presented.
Time Frame: Up to 2 years
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Participants
  Platelets transfusion | 5
  RBC transfusion | 4
  RBC concentrated transfusion | 1

33. Secondary Outcome: Part 2: Number of Participants With Any AEs and SAEs
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention or event associated with liver injury and impaired liver function were categorized as SAE.
Time Frame: Up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Part 2: Change From Baseline in Platelets, Neutrophils, Monocytes, Lymphocytes, Leucocyte, Eosinophils and Basophils at Indicated Time-points
Description: Blood samples were to be collected from participants for evaluation of hematology parameters including platelets, neutrophils, monocytes, lymphocytes, leucocyte, eosinophils and basophils. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Part 2: Change From Baseline in MCV at Indicated Time-points
Description: Blood samples were to be collected from participants for evaluation of hematology parameters including MCV. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Part 2: Change From Baseline in MCH at Indicated Time-points
Description: Blood samples were to be collected from participants for evaluation of hematology parameters including MCH. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Part 2: Change From Baseline in MCHC and Hb at Indicated Time-points
Description: Blood samples were to be collected from participants for evaluation of hematology parameters including MCHC and Hb. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Part 2: Change From Baseline in Hematocrit at Indicated Time-points
Description: Blood samples were to be collected from participants for evaluation of hematology parameters including Hematocrit. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Part 2: Change From Baseline in Erythrocytes at Indicated Time-points
Description: Blood samples were to be collected from participants for evaluation of hematology parameters including erythrocytes. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

40. Secondary Outcome: Part 2: Change From Baseline in Percent Reticulocytes at Indicated Time-points
Description: Blood samples were to be collected from participants for evaluation of hematology parameters including percent reticulocytes. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

41. Secondary Outcome: Part 2: Change From Baseline in Blast/Leukocytes at Indicated Time-points
Description: Blood samples were to be collected from participants for evaluation of hematology parameters including blast/leukocytes. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

42. Secondary Outcome: Part 2: Change From Baseline in ALT, ALP, AST, LDH and GGT at Indicated Time-points
Description: Blood samples were to be collected from participants for evaluation of clinical chemistry parameters including ALT, ALP, AST, LDH and GGT. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

43. Secondary Outcome: Part 2: Change From Baseline in Calcium, Chloride, Glucose, Potassium, Sodium, Phosphate and Urea Nitrogen at Indicated Time-points
Description: Blood samples were to be collected from participants for evaluation of clinical chemistry parameters including Calcium, chloride, glucose, potassium, sodium, phosphate and urea nitrogen. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

44. Secondary Outcome: Part 2: Change From Baseline in Total Bilirubin, Direct Bilirubin, Creatinine and Urate at Indicated Time Points
Description: Blood samples were to be collected from participants for evaluation of clinical chemistry parameters including Total Bilirubin, Direct Bilirubin, Creatinine and urate. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

45. Secondary Outcome: Part 2: Change From Baseline in Albumin and Protein at Indicated Time Points
Description: Blood samples were to be collected from participants for evaluation of clinical chemistry parameters including Albumin and Protein. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

46. Secondary Outcome: Part 2: Change From Baseline in pCO2 at Indicated Time Points
Description: Blood samples were to be collected from participants for evaluation of clinical chemistry parameters including pCO2. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

47. Secondary Outcome: Part 2: Change From Baseline in SBP and DBP at Indicated Time-points
Description: Vital signs including SBP and DBP were to be measured after resting for at least 5 minutes in a semi-supine position. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

48. Secondary Outcome: Part 2: Change From Baseline in Heart Rate at Indicated Time-points
Description: Vital signs including heart rate was to be measured after resting for at least 5 minutes in a semi-supine position. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

49. Secondary Outcome: Part 2: Change From Baseline in Respiratory Rate at Indicated Time-points
Description: Vital signs including respiratory rate was to be measured after resting for at least 5 minutes in a semi-supine position. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

50. Secondary Outcome: Part 2: Change From Baseline in Body Temperature at Indicated Time-points
Description: Vital signs including body temperature was to be measured after resting for at least 5 minutes in a semi-supine position. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

51. Secondary Outcome: Part 2: Change From Baseline in ECG Mean Heart Rate at Indicated Time-points
Description: Single 12-lead ECG was to be obtained at designated time points during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was to be calculated by subtracting post-dose value from Baseline value.
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

52. Secondary Outcome: Part 2: Change From Baseline in ECG PR Interval, QRS Duration, QT Interval, QTcB and QTcF at Indicated Time-points
Description: as for outcome 51
Time Frame: Baseline and up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

53. Secondary Outcome: Part 2: Number of Participants With Abnormal Findings During Physical Examination
Description: A complete physical examination included, at a minimum, assessment of the Cardiovascular, Respiratory, Gastrointestinal and Neurological systems. A brief physical examination included, at a minimum assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen).
Time Frame: Up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

54. Secondary Outcome: Part 2: Plasma Clearance (CL/F) of GSK2879552
Description: Blood samples were to be collected at indicated time points to evaluate CL/F of GSK2879552. Each PK sample was to be collected as close as possible to the planned time relative to the dose (i.e., time zero) administered to the participant on PK days.
Time Frame: Cycle 1, Day 1: pre-dose, 0.5, 1, 3 hour; pre-dose on Day 4; Day 7: pre-dose, 0.5, 1, 3 hour; Day 15: pre-dose, 0.5-1 hour post-dose; pre-dose on Day 22; Cycle 2: pre-dose on Days 1, 7, 15, 22; Pre-dose on Day 1 of Cycles 3 to 1 (each cycle of 28 days)
Population: PK Concentration Population. Data was not collected for this endpoint as study was terminated during Part 1 and Part 2 was not initiated.
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

55. Secondary Outcome: Part 2: Duration of Response
Description: Duration of response is defined as the time from first documented evidence of response until the first documented sign of disease progression or death. If no disease progression or death, the duration of response was to be censored at last disease assessment.
Time Frame: Up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

56. Secondary Outcome: Part 2: Progression-free Survival
Description: Progression-free survival is defined as the time from first treatment dose until the first documented sign of disease progression or death. If the participant missed more than one visit prior to the date of documented events, PFS was to be censored at the last adequate assessment prior to missing. Otherwise, if the participant did not have a documented date of events, PFS was to be censored at the date of the last adequate assessment.
Time Frame: Up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

57. Secondary Outcome: Part 2: Overall Survival
Description: Overall survival is defined as the time from first treatment dose until death due to any reason. For the analysis of overall survival, the last date of known contact was to be used for those participants who had not died at the time of analysis; such participants were to be considered censored.
Time Frame: Up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

58. Secondary Outcome: Part 2: Percentage of Participants With Disease Progression to AML
Description: The percentage of participants experiencing AML on the All Treated Subjects Population was to be presented.
Time Frame: Up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

59. Secondary Outcome: Part 2: Time to AML Progression
Description: Time to AML progression is defined as the time from first treatment dose until AML progression or crossover if using the All Treated Subjects Population. For the analysis of time to AML, if the participant did not experience AML, time to AML was to be censored at the last treatment prior to the initiation of anti-cancer therapy or crossover.
Time Frame: Up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

60. Secondary Outcome: Part 2: Number of Participants With Documented Platelet and Red Blood Cell (RBC) Transfusions Per Month
Description: Number of participants with documented platelet and RBC transfusions were to be presented.
Time Frame: Up to 2.5 years
Population: as for outcome 21
Arm/Group | Part 2: GSK2879552 | Part 2: GSK2879552+Azacitidine
Number analyzed (Participants) | 0 | 0

61. Primary Outcome: Part 1: Change From Baseline in Total Bilirubin, Direct Bilirubin, Creatinine and Urate at Indicated Time Points
Description: Blood samples were collected from participants for evaluation of clinical chemistry parameters including Total Bilirubin, Direct Bilirubin, Creatinine and urate. Baseline was defined as the value obtained prior to first dosing (Day 1). Change from Baseline was calculated by subtracting post-dose value from Baseline value.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Part 1: GSK2879552
Number analyzed (Participants) | 5
Micromoles per liter (umol/L)
  Total Bilirubin, Cycle 1, Day 1, n=4: number analyzed (Participants) | 4
  Total Bilirubin, Cycle 1, Day 1, n=4 | -3.420 (5.4075)
  Total Bilirubin Cycle 1, Day 7, n=5 | -1.094 (5.6580)
  Total Bilirubin Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Total Bilirubin Cycle 1, Day 15, n=4 | 0.128 (6.6278)
  Total Bilirubin Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Total Bilirubin Cycle 1, Day 22, n=3 | -1.710 (2.9618)
  Total Bilirubin Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Total Bilirubin Cycle 2, Day 1, n=3 | -2.850 (3.5596)
  Total Bilirubin Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Total Bilirubin Cycle 3, Day 1, n=3 | 0.000 (3.4200)
  Total Bilirubin Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Total Bilirubin Cycle 4, Day 1, n=2 | -0.855 (3.6275)
  Total Bilirubin, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Total Bilirubin, Cycle 5, Day 1, n=1 | -3.420 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Direct Bilirubin, Cycle 1, Day 1, n=1: number analyzed (Participants) | 1
  Direct Bilirubin, Cycle 1, Day 1, n=1 | 1.368 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Creatinine, Cycle 1, Day 1, n=4: number analyzed (Participants) | 4
  Creatinine, Cycle 1, Day 1, n=4 | 16.133 (25.5329)
  Creatinine Cycle 1, Day 7, n=5 | 4.066 (11.2271)
  Creatinine Cycle 1, Day 15, n=4: number analyzed (Participants) | 4
  Creatinine Cycle 1, Day 15, n=4 | 17.238 (17.4800)
  Creatinine Cycle 1, Day 22, n=3: number analyzed (Participants) | 3
  Creatinine Cycle 1, Day 22, n=3 | 23.279 (18.5500)
  Creatinine Cycle 2, Day 1, n=3: number analyzed (Participants) | 3
  Creatinine Cycle 2, Day 1, n=3 | 16.501 (16.6402)
  Creatinine Cycle 3, Day 1, n=3: number analyzed (Participants) | 3
  Creatinine Cycle 3, Day 1, n=3 | 15.912 (20.5613)
  Creatinine Cycle 4, Day 1, n=2: number analyzed (Participants) | 2
  Creatinine Cycle 4, Day 1, n=2 | 32.708 (8.7512)
  Creatinine, Cycle 5, Day 1, n=1: number analyzed (Participants) | 1
  Creatinine, Cycle 5, Day 1, n=1 | 4.420 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Urate, Cycle 1, Day 1, n=1: number analyzed (Participants) | 1
  Urate, Cycle 1, Day 1, n=1 | 41.636 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Urate Cycle 1, Day 7, n=2: number analyzed (Participants) | 2
  Urate Cycle 1, Day 7, n=2 | 5.948 (0.0000)
  Urate Cycle 1, Day 22, n=1: number analyzed (Participants) | 1
  Urate Cycle 1, Day 22, n=1 | 35.688 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Urate Cycle 2, Day 1, n=1: number analyzed (Participants) | 1
  Urate Cycle 2, Day 1, n=1 | 65.428 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Urate Cycle 3, Day 1, n=1: number analyzed (Participants) | 1
  Urate Cycle 3, Day 1, n=1 | 89.220 (NA) — Standard deviation could not be calculated due to insufficient number of participants.
  Urate Cycle 4, Day 1, n=1: number analyzed (Participants) | 1
  Urate Cycle 4, Day 1, n=1 | 59.480 (NA) — Standard deviation could not be calculated due to insufficient number of participants.

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and Non-serious adverse events (Non-SAEs) were collected from the start of the study treatment up to Cycle 5 (each cycle of 28 days) in Part 1.
Description: SAEs and Non-SAEs were reported by treatment for the All Treated Subjects Population which comprised of all participants who received at least one dose of study treatment. Data is presented for Part 1 only as data was not collected in Part 2 due to the study was terminated during Part 1 only, and Part 2 was not initiated.
Arm/Group | Part 1: GSK2879552
All-Cause Mortality (participants affected / at risk) | 2/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: GSK2879552 (N=5)
Sinusitis (Infections and infestations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: GSK2879552 (N=5)
Fatigue (General disorders) | 3
Oedema (General disorders) | 1
Pyrexia (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Balance disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Parosmia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Blood blister (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Fungal infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT02929498/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT02929498/SAP_001.pdf